CLINICAL TRIAL: NCT00684866
Title: A Cumulative Dose Tolerability Study of Levalbuterol HFA and Racemic Albuterol HFA in Pediatric Subjects With Asthma
Brief Title: Safety and Tolerability Study of Levalbuterol HFA and Racemic Albuterol HFA in Pediatrics Subjects With Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 051-311
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Asthma
Keywords: Asthma; Levalbuterol; Racemic Albuterol
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Subjects will receive both treatments: (a) levalbuterol HFA MDI; 45 micrograms (8 cumulative doses); followed by (b) racemic albuterol HFA MDI; 90 micrograms (8 cumulative doses).
  The first treatment will be administered, followed by a 7 ±2 days washout period, after which the second of the two treatments will be administered. Cumulative dosing will occur according to the following schedule: 1 puff at 0 and 30 minutes, 2 puffs at 60 minutes, 4 puffs at 90 minutes and 8 puffs at 120 minutes. Treatment will be administered with an AeroChamber Plus ™ spacer for the first cohort (spacer cohort) of subjects and without the AeroChamber Plus ™ spacer (non-spacer cohort) for the second cohort of subjects.
  Interventions: Drug: Levalbuterol HFA MDI followed by Racemic albuterol HFA MDI
- B (Active Comparator): Subjects will receive both treatments: (a) racemic albuterol HFA MDI; 90 micrograms (16 cumulative doses) followed by (b) levalbuterol HFA MDI; 45 micrograms (16 cumulative doses) The first treatment will be administered, followed by a 7 ±2 days washout period, after which the second of the two treatments will be administered. Cumulative dosing will occur according to the following schedule: 1 puff at 0 and 30 minutes, 2 puffs at 60 minutes, 4 puffs at 90 minutes and 8 puffs at 120 minutes. Treatment will be administered with an AeroChamber Plus ™ spacer for the first cohort (spacer cohort) of subjects and without the AeroChamber Plus ™ spacer (non-spacer cohort) for the second cohort of subjects.
  Interventions: Drug: Racemic Albuterol followed by levalbuterol HFA MDI

INTERVENTIONS:
Drug: Levalbuterol HFA MDI followed by Racemic albuterol HFA MDI — (a) Subjects will receive both treatments: (a) levalbuterol HFA MDI; 45 micrograms (16 cumulative doses); followed by (b) racemic albuterol HFA MDI; 90 micrograms (16 cumulative doses)
  Other Names: Xopenex HFA MDI; albuterol HFA MDI
  Arms: A
Drug: Racemic Albuterol followed by levalbuterol HFA MDI — (a) Subjects will receive both treatments: (a) racemic albuterol HFA MDI; 90 micrograms (16 cumulative doses) followed by (b) levalbuterol HFA MDI; 45 micrograms (16 cumulative doses)
  Other Names: albuterol HFA MDI; Xopenex HFA MDI
  Arms: B

SUMMARY:
The purpose of this study is to compare the safety and tolerability of levalbuterol HFA metered dose inhaler (MDI) versus racemic albuterol HFA MDI in pediatric subjects 4-11 years of age with asthma

DETAILED DESCRIPTION:
A randomized, double-blind, active-controlled multicenter, two-way crossover study of HFA levalbuterol (with and without a spacer) in subjects 4-11 years of age with asthma. This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria:

* Subject, male or female, must be between the ages of 4 to 11 years, inclusive, at the time of consent.
* Female subjects who are 8 years of age or older will have a negative serum pregnancy test at study start.
* Subject must have a documented diagnosis of asthma for a minimum of 6 months prior to study start.
* Subject must be in good health with the exception of their reversible airways disease and not suffering from any chronic condition that might affect their respiratory function.
* Subject must have a chest X-ray or have one taken within 12 months prior to randomization may be used.
* Subject's parent/legal guardian must be able to complete the diary cards and medical event calendars reliably on a daily basis and understand dosing instructions. Any subject who is not able to do this must have a parent/legal guardian who can assist them during the study with these activities.

Exclusion Criteria:

* Female subject who is pregnant or lactating.
* Subject who has participated in an investigational drug study within 30 days prior to study start, or who is currently participating in another clinical trial.
* Subject whose schedule prevents him or her from taking the first daily dose of study medication and/or starting study visits before 9 AM.
* Subject who has travel commitments during the study that would interfere with trial measurements or compliance or both.
* Subject who has a history of hospitalization for asthma within 4 weeks prior to study start, or who is scheduled for in-patient hospitalization, including elective surgery during the course of the trial
* Subject with a known sensitivity to levalbuterol or racemic albuterol, or any of the excipients contained in any of these formulations.
* Subject using any prescription drug with which albuterol sulfate administration is contraindicated.
* Subject with currently diagnosed life-threatening asthma defined as a history of asthma episodes requiring intubation, associated with hypercapnia, respiratory arrest, or hypoxic seizures within 3 months prior to study start.
* Subject with a history of cancer.
* Subject with hyperthyroidism, diabetes, hypertension, cardiac diseases or seizure disorders.
* Subject with a history of substance abuse or drug abuse within 12 months preceding study start.
* Subject with a history of cigarette smoking or use of any tobacco products.
* Subject with a documented history of bronchopulmonary aspergillosis or any form of allergic alveolitis.
* Subject who has suffered from a clinically significant upper or lower respiratory tract infection in the 2 weeks prior to study start.
* Subject with unstable asthma; or who have had a change in asthma therapy; or a visit to the Emergency Department or hospital for worsening asthma within 4 weeks.
* Subject who is a staff member or relative of a staff member.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2003-01; Primary Completion 2003-07 (Actual); Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Increases from visit pre-dose to each post-dose dose measurement in heart rate, blood pressure (systolic and diastolic), potassium and glucose | 0, 7, 10 days

SECONDARY OUTCOMES:
Percent change in FEV1 (from visit pre-dose to each post dose measure) | Days 0, 7, 10
Percent change in FVC (from visit pre-dose to each post dose measure) | Days 0, 7, 10
Percent change in FEF25-75% (from visit pre-dose to each post dose measure) | Days 0, 7, 10
Number of cumulative actuations received | Days 0, 7, 10

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Madera, California
  - San Diego, California
  - Savannah, Georgia
  - Louisville, Kentucky
  - Cortland, New York
  - Medford, Oregon
  - Portland, Oregon
  - Chester, Pennsylvania
  - Knoxville, Tennessee
  - Dallas, Texas
  - Houston, Texas